CLINICAL TRIAL: NCT00366639
Title: ADHERE Core III - Acute Decompensated Heart Failure Registry
Brief Title: Registry for Acute Decompensated Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: Scios, Inc. (Industry)
Responsible Party: Sr. Director, Clinical Team Leader, Scios
Other Study IDs: CR005194; NCT00530673 (obsolete NCT alias)
Record Dates: First submitted 2006-08-18; First posted 2006-08-21 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Heart Failure, Congestive; Heart Decompensation
Keywords: Heart failure, congestive; Heart decompensation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 001
  Interventions: Other: Acute Decompensated Heart Failure

INTERVENTIONS:
Other: Acute Decompensated Heart Failure — Treatment & outcomes during hospital admission for Acute DHF

SUMMARY:
The purpose of the ADHERE study is to develop a multi-center, observational, open-label registry of the management strategies of patients treated in the hospital for acute Heart Failure in the United States.

DETAILED DESCRIPTION:
The objective is to compile a clinical database on the strategy for the medical management of patients hospitalized with acute Heart Failure (HF). Through the use of the information collected from acute care hospitals across the United States the following information may be coming out of this study: 1) Assist hospitals in evaluating and improving quality of care for patients with acute HF by tracking quality indicators and providing benchmark data reports; 2) Describe the demographic and clinical characteristics of patients who are hospitalized with acute HF; 3) Characterize the initial emergency department evaluation and subsequent inpatient management of patients hospitalized with acute HF; 4) Identify patient characteristics and medical care practices associated with improved health outcomes in those hospitalized with acute HF; 5) Characterize trends and changes over time in the management of acute HF; 6) Offer surveillance of adherence to practice guidelines as these emerge for the inpatient management of acute HF. Observational Study - No investigational drug administered

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years at the time of admission to the hospital
* Received or is eligible to receive a principal hospital discharge diagnosis of HF
* Decompensated HF is present as determined clinically by the patient care team

Exclusion Criteria:

* HF is present as a co-morbid condition, but is not a principal focus of diagnosis or treatment during this hospitalization episode

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients admitted to an acute care hospital and treated actively for acute HF, where acute HF is defined clinically as a new onset with HF decompensation
Sampling Method: Non-Probability Sample
Enrollment: 24118 (Actual)
Dates: Start 2001-10; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Course of care in the Emergency Department (ED) and course of care in the inpatient hospital, use of diuretics (increase urine excretion) vasodilators (relax artey and veins) and inotropeic agents (increase the function of the heart) rate of death | From admission to discharge from the hospital

SECONDARY OUTCOMES:
Data from patient demographics ( sex, age, gender, race) | at patients admission

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.

REFERENCES:
- [Derived] Kociol RD, Hammill BG, Fonarow GC, Klaskala W, Mills RM, Hernandez AF, Curtis LH. Generalizability and longitudinal outcomes of a national heart failure clinical registry: Comparison of Acute Decompensated Heart Failure National Registry (ADHERE) and non-ADHERE Medicare beneficiaries. Am Heart J. 2010 Nov;160(5):885-92. doi: 10.1016/j.ahj.2010.07.020. PMID 21095276
- [Derived] Maisel AS, Peacock WF, McMullin N, Jessie R, Fonarow GC, Wynne J, Mills RM. Timing of immunoreactive B-type natriuretic peptide levels and treatment delay in acute decompensated heart failure: an ADHERE (Acute Decompensated Heart Failure National Registry) analysis. J Am Coll Cardiol. 2008 Aug 12;52(7):534-40. doi: 10.1016/j.jacc.2008.05.010. PMID 18687247
- [Derived] Kamath SA, Drazner MH, Wynne J, Fonarow GC, Yancy CW. Characteristics and outcomes in African American patients with decompensated heart failure. Arch Intern Med. 2008 Jun 9;168(11):1152-8. doi: 10.1001/archinte.168.11.1152. PMID 18541822
- [Derived] Peacock WF 4th, De Marco T, Fonarow GC, Diercks D, Wynne J, Apple FS, Wu AH; ADHERE Investigators. Cardiac troponin and outcome in acute heart failure. N Engl J Med. 2008 May 15;358(20):2117-26. doi: 10.1056/NEJMoa0706824. PMID 18480204
- [Derived] Fonarow GC, Peacock WF, Horwich TB, Phillips CO, Givertz MM, Lopatin M, Wynne J; ADHERE Scientific Advisory Committee and Investigators. Usefulness of B-type natriuretic peptide and cardiac troponin levels to predict in-hospital mortality from ADHERE. Am J Cardiol. 2008 Jan 15;101(2):231-7. doi: 10.1016/j.amjcard.2007.07.066. Epub 2007 Dec 3. PMID 18178412
- [Derived] Hauptman PJ, Goodlin SJ, Lopatin M, Costanzo MR, Fonarow GC, Yancy CW. Characteristics of patients hospitalized with acute decompensated heart failure who are referred for hospice care. Arch Intern Med. 2007 Oct 8;167(18):1990-7. doi: 10.1001/archinte.167.18.1990. PMID 17923600
- [Derived] Fonarow GC, Peacock WF, Phillips CO, Givertz MM, Lopatin M; ADHERE Scientific Advisory Committee and Investigators. Admission B-type natriuretic peptide levels and in-hospital mortality in acute decompensated heart failure. J Am Coll Cardiol. 2007 May 15;49(19):1943-50. doi: 10.1016/j.jacc.2007.02.037. Epub 2007 Apr 30. PMID 17498579